CLINICAL TRIAL: NCT05729152
Title: LONGCOVID WP3 "Cardiovascular Events for a Long Time End of COVID 19 Infection "
Brief Title: Cardiovascular Events for a Long Time End of COVID 19 Infection
Acronym: LONGCOVIDWP3
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Pedicino Daniela, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5031
Record Dates: First submitted 2023-02-13; First posted 2023-02-15 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Myocardial Disease
Keywords: acute myocardial injury; COVID-19
MeSH Terms: conditions — Cardiomyopathies; COVID-19 | interventions — epicatechin gallate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sample blood — Partecipants will undergo a baseline assessment by history, objective examination, laboratory tests, ECG, 6-minute walking test and echocardiogram
  Other Names: Objective examination, laboratory tests, ECG, 6-minute walking test and echocardiogram

SUMMARY:
In the follow-up of partecipants with Covid-19 infection, persistence of cardiovascular symptoms is common. Studies on the acute phase of Covid-19 infection have demonstrated a significant prevalence of acute myocardial damage (15-44%), and imaging studies have confirmed the presence of structural changes in the pericardium and myocardium several months after the acute phase. The aim of the project is to identify the prevalence and characteristics of long-term cardiovascular changes in Covid-19 infection.

DETAILED DESCRIPTION:
The study is a continuation of the "CARDICoVRISK" registry project ("Cardiovascular risk and effects ancillary effects of cardiology drug therapy during n-CoV-19 infection"), which collected data on alterations cardiovascular changes during the acute phase and shortly after the acute phase.

The design of the current study is observational cross-sectional comparison with historical data. The study plans to enroll 240 patients hospitalized during the acute phase of COVID-19 infection. Enrollment of patients will be carried out in three separate centers. Enrolled patients will undergo a baseline assessment by history, objective examination, laboratory tests, ECG, 6-minute walking test and echocardiogram.

ELIGIBILITY:
Inclusion Criteria:

* partecipants with previous hospitalization for Covid-19 infection confirmed by pharyngeal molecular swab at least 12 months prior to enrollment;
* adult partecipants between the ages of 18 and 90 years old;
* signature of informed consent;

Exclusion Criteria:

* partecipants with poor echocardiographic acoustic window impairing the performance of the examination
* partecipants with atrial fibrillation
* partecipants with ischemic or nonischemic heart disease with known decreased systolic function of the left ventricle left

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study plans to enroll 240 partecipants hospitalized during the acute phase of COVID-19 infection.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2023-05-26 (Estimated)

PRIMARY OUTCOMES:
Identify long-term myocardial damage and compare it with the prevalence and extent of acute myocardial damage in approximately 240 subjects who have been affected by COVID 19 | 6 months
  The main purpose of this study is to identify long-term myocardial damage and compare it with the prevalence and extent of acute myocardial damage. The anatomical and functional substrates of cardiovascular manifestations will be analyzed by basic and advanced echocardiographic technologies and, when appropriate, by MRI cardiac magnetic resonance imaging.
  Acute myocardial damage will be estimated by observation of troponin values already collected during acute infection as part of the CARDICoVRISK registry. Distant myocardial damage will be assessed by the assessments provided in the baseline visit.

SECONDARY OUTCOMES:
Evaluate functional and anatomical abnormalities on diastolic dysfunction in 240 subjects who reported cardiac abnormalities following Covid infection | 3 months
  A secondary objective is to evaluate functional and anatomical abnormalities as pathophysiologic substrates of dysfunction diastolic and the onset of heart failure at preserved ejection fraction, furthermore in partecipants who, during the baseline visit, will show cardiac alterations the execution of a cardiac magnetic resonance examination will be evaluated.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Istituto Auxologico Italiano IRCSS Ospedale San Luca, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma